CLINICAL TRIAL: NCT06526468
Title: CHinese pulmOnary Embolism Multimodality Imaging-artifiCial intelligencE Study
Brief Title: Chinese PE Multimodality Imaging Artificial Intelligence Study
Status: Recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Clinical Professor, China-Japan Friendship Hospital
Other Study IDs: CHOICE
Record Dates: First submitted 2024-06-15; First posted 2024-07-29 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Embolism; Chronic Thromboembolic Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Disease
Keywords: imaging; early diagnosis; differential diagnosis; risk stratification; prognosis assessment
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and PEA specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute pulmonary embolism cohort: 1. Patients objectively confirmed acute symptomatic PE or PE with deep vein thrombosis (DVT)
  2. PE was confirmed by CTPA, lung V/Q scan or pulmonary angiography.
  Interventions: Device: Artificial Intelligence
- Chronic thromboembolic pulmonary disease without pulmonary hypertension cohort: 1. Patients with functional impairment despite 3 months of adequate anticoagulation therapy after APE.
  2. CTPA/ pulmonary angiography or V/Q scan showed unresolved thrombi in the pulmonary vessels.
  3. Without pulmonary hypertension at rest(mean pulmonary arterial pressure (mPAP) <20 mmHg), as measured by right heart catheterization.
  Interventions: Device: Artificial Intelligence
- Chronic thromboembolic pulmonary hypertension cohort: 1. Patients with functional impairment despite 3 months of adequate anticoagulation therapy
  2. CTPA/ pulmonary angiography or V/Q scan showed unresolved thrombi in the pulmonary vessels.
  3. With pulmonary hypertension at rest (mean pulmonary arterial pressure (mPAP) >20 mmHg), as measured by right heart catheterization.
  Interventions: Device: Artificial Intelligence
- Other pulmonary vascular disease cohort: Patients diagnosed with other pulmonary vascular disease including Takayasu arteritis, pulmonary artery sarcoma, and fibrosing mediastinitis.
  Interventions: Device: Artificial Intelligence

INTERVENTIONS:
Device: Artificial Intelligence — AI technology will provide novel imaging markers and generate a radiology report with relevant key slice imaging and evaluation results

SUMMARY:
The CHinese pulmOnary Embolism Multimodality Imaging-artifiCial intelligencE Study (CHOICE) is a prospective observational multi-center study that will collect imaging text data and raw data of patients with pulmonary embolism (PE) in China. By combining artificial intelligence technology, it aims to identify imaging markers to assist in early diagnosis, differential diagnosis, risk stratification, and prognosis assessment of PE.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) represents a significant public health issue. Timely diagnosis and treatment during the acute phase, as well as appropriate long-term follow-up strategies, are crucial for the management of PE. PE is classified into three stages based on disease course: acute pulmonary embolism (APE), chronic thromboembolic pulmonary disease (CTEPD), and chronic thromboembolic pulmonary hypertension (CTEPH). APE can cause acute right ventricular failure and death if not diagnosed and treated early. CTEPD has the potential to significantly impair patients' quality of life. CTEPH is a rare and potentially life-threatening long-term sequelae of PE, characterized by persistent obstruction of pulmonary arteries by organized clots, leading to redistribution of blood flow and secondary remodeling of the pulmonary microvasculature. Early identification of PE and implementation of targeted treatment plans will significantly improve survival rates and prognosis.

Multimodal imaging tests play a crucial role in the management of PE (including computed tomography pulmonary angiography (CTPA), magnetic resonance imaging (MRI), echocardiography, and lung ventilation/perfusion (V/Q) scan). The guidelines have identified the right ventricle to left ventricle (RV:LV) ratio >1.0 on CTPA or right heart dysfunction signs from echocardiography as important indicators for risk stratification of APE. Patients stratified as high risk require closer monitoring in an inpatient setting. Whereas, those stratified as low risk are suitable for early discharge.

Therefore, exploring novel imaging markers and integrating these markers into radiology reports may have potential clinical significance. If no quantifiable evidence of right ventricular dysfunction is provided to clinicians to make treatment decisions, patients with high-risk APE may be considered "low-risk" and discharged home. In addition, patients with low-risk APE may require longer hospital stays and may not need to be hospitalized, which undoubtedly increases healthcare costs. For patients with CTEPD or CTEPH, treatment options are diverse, including multimodal therapies such as pulmonary endarterectomy, balloon pulmonary angioplasty and targeted medical therapy. Therefore, multimodal imaging evaluation is meaningful for clinical treatment decision-making and efficacy monitoring. Combined with artificial intelligence (AI) technology, it can provide a variety of metrics to assist in evaluating clots morphology, pulmonary ventilation-perfusion function, cardiac function, hemodynamics, and more. AI can not only assist in finding more clinically significant imaging biomarkers but also customize standardized radiology reports, which are expected to address the current challenges.

This study is a multi-center real-world study aimed at exploring novel imaging markers in combination with AI technology and integrating them into a software for clinical application to provide quantitative parameters, using imaging reports and raw data from Chinese patients with PE. It is hypothesized that AI technology can improve early diagnosis, differential diagnosis, risk stratification, and management of PE by increasing the ability to accurately evaluate PE in a real-world clinical setting. The researchers also hypothesized that the integration of AI technologies would be cost-effective and acceptable to radiologists and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* 14 Years and older
* Patients suspected of PE

Exclusion Criteria:

* Pregnant women
* Refuse to follow up
* Incomplete or discontinued imaging scans
* Insufficient quality of image data to allow for analysis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected of PE in China
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of PE | 2 years
  Comparison before and after AI technique.
APE risk stratification rates (low, intermediate low, intermediate high and high risk) | 2 years
  Comparison before and after AI technique.
Disease severity of chronic thromboembolic pulmonary disease (CTEPD)/chronic thromboembolic pulmonary hypertension (CTEPH) | 2 years
  Comparison before and after AI technique. Assessment of disease severity is comprehensive, referring to the comprehensive risk assessment in pulmonary arterial hypertension (three-strata model) [DOI: 10.1183/13993003.00879-2022], including clinical observations and modiﬁable variables. The higher the score, the more severe the condition.
30 day mortality | 2 years
  Patient mortality (death) at 30-days post-PE diagnosis. Comparison before and after AI technique.

SECONDARY OUTCOMES:
Rate of discordant PE cases | 2 years
  False positive and false negative rate
AI failure rate for PE detection | 2 years
  Proportion of scans unable to be interpreted by AI despite suitable CTPA acquisition
12 month mortality | 2 years
  Patient mortality (death) at 12-months post-PE diagnosis. Comparison before and after AI technique.
Length of hospital stay for PE | 2 years
  Comparison before and after AI technique. Measured as number of days from admission to time of discharge from hospital.
Time from symptom onset to final diagnosis | 3 months
  Comparison before and after AI technique.
Hospitalization cost for PE using Markov model | 2 years
  Comparison before and after AI technique.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, PhD, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Frendship hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Information gathered for this study will not be disclosed to any other person or entity, or for other research.

REFERENCES:
- [Derived] Xi L, Wang J, Liu A, Ni Y, Du J, Huang Q, Li Y, Wen J, Wang H, Zhang S, Zhang Y, Zhang Z, Wang D, Xie W, Gao Q, Cheng Y, Zhai Z, Liu M. Development of a lung perfusion automated quantitative model based on dual-energy CT pulmonary angiography in patients with chronic pulmonary thromboembolism. Insights Imaging. 2025 Aug 18;16(1):182. doi: 10.1186/s13244-025-02067-6. PMID 40825922